CLINICAL TRIAL: NCT00661999
Title: A Phase III, Randomized Study of the Effects of Parenteral Iron, Oral Iron, or No Iron Supplementation on the Erythropoietic Response to Darbepoetin Alfa for Cancer Patients With Chemotherapy-Associated Anemia
Brief Title: Darbepoetin Alfa With or Without Iron in Treating Anemia Caused By Chemotherapy in Patients With Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Charles Lawrence Loprinzi, M.D., Mayo Clinic Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CDR0000593480; P30CA015083 (NIH); MC04CC (Other: Mayo Clinic Cancer Center); NCI-2009-01226 (Registry Identifier: NCI-CTRP); 1713-05 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2008-04-18; First posted 2008-04-21 (Estimated); Results first posted 2011-04-18 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-05

CONDITIONS: Anemia; Leukemia; Lymphoma; Lymphoproliferative Disorder; Multiple Myeloma and Plasma Cell Neoplasm; Precancerous Condition; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; monoclonal gammopathy of undetermined significance; extramedullary plasmacytoma; isolated plasmacytoma of bone; refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; primary systemic amyloidosis; Waldenstrom macroglobulinemia; post-transplant lymphoproliferative disorder; stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult grade III lymphomatoid granulomatosis; stage I adult Burkitt lymphoma; stage III adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult lymphoblastic lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; stage I adult diffuse large cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage III adult lymphoblastic lymphoma; stage IV adult lymphoblastic lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage I mantle cell lymphoma; stage I marginal zone lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; adult acute lymphoblastic leukemia in remission; recurrent adult acute lymphoblastic leukemia; untreated adult acute lymphoblastic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; progressive hairy cell leukemia, initial treatment; prolymphocytic leukemia; anemia; T-cell large granular lymphocyte leukemia; acute undifferentiated leukemia; mast cell leukemia; adult nasal type extranodal NK/T-cell lymphoma; untreated hairy cell leukemia
MeSH Terms: conditions — Anemia; Leukemia; Lymphoma; Lymphoproliferative Disorders; Multiple Myeloma; Neoplasms, Plasma Cell; Precancerous Conditions; Monoclonal Gammopathy of Undetermined Significance; Immunoglobulin Light-chain Amyloidosis; Waldenstrom Macroglobulinemia; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Hodgkin Disease; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Leukemia, Prolymphocytic; Leukemia, Large Granular Lymphocytic; Leukemia, Biphenotypic, Acute; Leukemia, Mast-Cell; Lymphoma, Extranodal NK-T-Cell | interventions — Darbepoetin alfa; ferrous sulfate; ferric gluconate; Sucrose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (Experimental): Patients receive darbepoetin alfa subcutaneously and sodium ferric gluconate complex IV over 90 minutes on day 1. Treatment repeats every 21 days for up to 15 weeks in the absence of unacceptable toxicity.
  Interventions: Biological: darbepoetin alfa; Drug: sodium ferric gluconate complex in sucrose
- Arm II (Experimental): Patients receive darbepoetin alfa as in arm I and oral ferrous sulfate once daily on days 1-21. Treatment repeats every 21 days for up to 15 weeks in the absence of unacceptable toxicity.
  Interventions: Biological: darbepoetin alfa; Dietary Supplement: ferrous sulfate
- Arm III (Experimental): Patients receive darbepoetin alfa as in arm I and oral placebo once daily on days 1-21. Treatment repeats every 21 days for up to 15 weeks in the absence of unacceptable toxicity.
  Interventions: Biological: darbepoetin alfa; Other: placebo

INTERVENTIONS:
Biological: darbepoetin alfa — Given by injection
Dietary Supplement: ferrous sulfate — Given by mouth
  Arms: Arm II
Drug: sodium ferric gluconate complex in sucrose — Given by IV
  Arms: Arm I
Other: placebo — Given by mouth
  Arms: Arm III

SUMMARY:
RATIONALE: Darbepoetin alfa may cause the body to make more red blood cells. Red blood cells contain iron that is needed to carry oxygen to the tissues. It is not yet known whether giving darbepoetin alfa (DA) together with intravenous iron or oral iron is more effective than giving darbepoetin alfa together with a placebo in treating anemia caused by chemotherapy.

PURPOSE: This randomized phase III trial is studying giving darbepoetin alfa together with iron to see how well it works compared with giving darbepoetin alfa together with a placebo in treating anemia caused by chemotherapy in patients with cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the effects of IV iron, oral iron, or placebo in combination with darbepoetin alfa on the hematopoietic response rate, defined as a hemoglobin increment of ≥ 2.0 g/dL from baseline or achievement of hemoglobin of ≥ 11 g/dL in the absence of red blood cell transfusions (RBC) in the preceding 28 days of the treatment period, in cancer patients with chemotherapy-associated anemia.

Secondary

* To compare the effects of these regimens on the mean hemoglobin increment from baseline to weeks 7 and 16 in these patients.
* To compare the effects of these regimens on the percentage of patients maintaining an average hemoglobin level within the American Society of Hematology/American Society of Clinical Oncology (ASH/ASCO)and National Comprehensive Cancer Network(NCCN) guideline-based target hemoglobin range (11-13 g/dL), once achieving a hemoglobin of ≥ 11 g/dL from week 1 to week 16 in the absence of RBC transfusions in the preceding 28 days of the treatment period.
* To compare the effects of intravenously (IV) iron, oral iron, or placebo on the response to darbepoetin alfa, in terms of time to achieving hemoglobin levels of ≥ 11g/dL.
* To compare the effects of these regimens on the percentage of patients who require RBC transfusions and the total transfusion needs.
* To compare the effects of these regimens on the change in hemoglobin week by week.
* To compare the effects of these regimens on quality-of-life changes from baseline to weeks 7 and 16.
* To identify if patients with inflammation (as indicated by elevated C-reactive protein (CRP) and serum hepcidin levels or low soluble transferrin receptor (sTfR)/log ferritin ratios) respond differently to darbepoetin alfa and iron therapy than patients without inflammation.

OUTLINE: Patients are stratified according to severity of anemia (mild [hemoglobin ≥ 9.5 g/dL] vs severe [hemoglobin < 9.5 g/dL]), treatment with a platinum-containing regimen (yes vs no), and gender. Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive darbepoetin alfa subcutaneously and sodium ferric gluconate complex IV over 90 minutes on day 1.
* Arm II: Patients receive darbepoetin alfa as in arm I and oral ferrous sulfate once daily on days 1-21.
* Arm III: Patients receive darbepoetin alfa as in arm I and oral placebo once daily on days 1-21.

In all arms, treatment repeats every 21 days for up to 15 weeks in the absence of unacceptable toxicity.

Patients complete quality-of-life (QOL) questionnaires in weeks 1, 7, and 16.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of a non-myeloid cancer (other than non-melanomatous skin cancer)
* Receiving or scheduled to receive chemotherapy (biological agents, such as small molecules/tyrosine kinase inhibitors and antibody-based therapies, are allowed)
* Has chemotherapy-related anemia (hemoglobin < 11 g/dL)

  * No anemia known to be secondary to gastrointestinal bleeding or hemolysis
  * No anemia known to be secondary to vitamin B12 or folic acid deficiency

    + Vitamin B12 and folic acid deficiency must be ruled out if the mean corpuscular volume (MCV) is > 100 fL
  * No anemia secondary to chemotherapy-induced myelodysplastic syndromes
* No primary hematologic disorder causing moderate to severe anemia (e.g., congenital dyserythropoietic anemia, homozygous hemoglobin S disease or compound heterozygous sickling states, or thalassemia major)

  - Carriers for these disease states are eligible
* No first-degree relative with primary hemochromatosis (unless the patient has undergone HFE genotyping and was found to have at least one wild-type allele, while the proband in the family demonstrated to have either the common C282Y or H63D mutation)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Ferritin > 20 mcg/L (i.e., not obviously iron deficient)
* ALT or AST < 5 times upper limit of normal
* Alert, mentally competent, and able to sign informed consent
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* Willing or able to be randomized and undergo study treatment
* Willing or able to fill out quality-of-life forms
* No uncontrolled hypertension (i.e., systolic blood pressure [BP] ≥ 180 mm Hg or diastolic BP ≥ 100 mm Hg)
* No history of uncontrolled cardiac arrhythmias
* No pulmonary embolism or deep venous thrombosis within the past year (unless the patient is on anticoagulation therapy and planning to continue it during study participation)
* No known hypersensitivity to darbepoetin alfa, erythropoietin, mammalian cell-derived products, iron, or human albumin
* No seizures within the past 3 months
* No gastrointestinal conditions expected to cause significant impairment of oral iron, such as untreated celiac disease or amyloidosis involving the gut - Patients with celiac disease who are adhering to a gluten-free diet are eligible

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 3 months since prior darbepoetin alfa, epoetin alfa, or any investigational forms of erythropoietin (e.g., gene-activated erythropoietin or novel erythropoiesis-stimulating protein)
* More than 1 year since prior peripheral blood stem cell or bone marrow transplantation
* More than 2 weeks since prior red blood cell transfusions
* More than 14 days since prior major surgery
* No prior gastrectomy or resection of > 100 cm of small intestine
* Not planning to undergo stem cell or bone marrow transplantation within the next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2006-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles L. Loprinzi, MD, Study Chair — Mayo Clinic; Tom R. Fitch, M.D., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Five-hundred and two (502) participants were recruited between February 2006 and December 2008 at Mayo Clinic Cancer Research Consortium (MCCRC) sites.
Pre-assignment Details: Eight patients canceled before the first dose of darbepoetin alfa (DA) (3 DA + Intravenously (IV) Iron, 3 DA + Oral Iron and 2 DA + Placebo); and 4 patients were ineligible (2 DA + Oral Iron, 2 DA + Placebo). These 12 patients were excluded from all analysis.
Groups:
- DA + IV Iron: Patients receive darbepoetin alfa (DA) subcutaneously and sodium ferric gluconate complex intravenously (IV) over 90 minutes on day 1. Treatment repeats every 21 days for up to 15 weeks in the absence of unacceptable toxicity.
- DA + Oral Iron: Patients receive darbepoetin alfa (DA) as in arm I and oral ferrous sulfate once daily on days 1-21. Treatment repeats every 21 days for up to 15 weeks in the absence of unacceptable toxicity.
- DA + Placebo: Patients receive darbepoetin alfa (DA) as in arm I and oral placebo once daily on days 1-21. Treatment repeats every 21 days for up to 15 weeks in the absence of unacceptable toxicity.
Period: Overall Study
Arm/Group | DA + IV Iron | DA + Oral Iron | DA + Placebo
Started | 164 | 163 | 163
Completed | 105 | 113 | 106
Not Completed | 59 | 50 | 57
Not completed — Adverse Event | 11 | 5 | 8
Not completed — Death | 8 | 6 | 3
Not completed — Other Reasons | 5 | 12 | 23
Not completed — Withdrawal by Subject | 30 | 23 | 14
Not completed — Alternative Treatment | 1 | 0 | 0
Not completed — Other Medical Problems | 4 | 4 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DA + IV Iron | DA + Oral Iron | DA + Placebo | Total
Number analyzed (Participants) | 164 | 163 | 163 | 490
Age Continuous [Mean (Standard Deviation); unit: years] | 64 (11) | 63 (13) | 63 (11) | 63 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 106 | 105 | 320
  Male | 55 | 57 | 58 | 170
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 1 | 4
  Asian | 0 | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 7 | 4 | 17
  White | 155 | 147 | 156 | 458
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 1 | 7
Degree of Anemia [Number; unit: Participants]
  Mild: Hemoglobin>=9.5 | 123 | 123 | 123 | 369
  Severe: Hemoglobin <9.5 | 41 | 40 | 40 | 121
Platinum-Containing Regimen [Number; unit: Participants]
  Yes | 79 | 79 | 78 | 236
  No | 85 | 84 | 85 | 254
Tumor Type [Number; unit: Participants]
  Hematologic Neoplasm | 6 | 8 | 11 | 25
  Solid Tumor | 157 | 154 | 151 | 462
  Both | 1 | 1 | 1 | 3
Weight [Mean (Standard Deviation); unit: kg] | 77.4 (18.74) | 79.4 (19.75) | 76.4 (17.68) | 77.7 (18.75)
Height [Mean (Standard Deviation); unit: cm] | 166.9 (9.44) | 167.7 (8.93) | 166.8 (9.36) | 167.1 (9.24)
Baseline Ferritin [Mean (Standard Deviation); unit: µg/L] | 460.5 (526.99) | 479.5 (484.15) | 456.0 (479.27) | 465.3 (496.41)
Baseline Transferrin Saturation [Mean (Standard Deviation); unit: Percentage Saturation] | 22.5 (12.81) | 19.6 (11.7) | 22.2 (13.36) | 21.5 (12.69)

OUTCOME MEASURES:

1. Primary Outcome: Hematopoietic Response Rate Defined as the Number of Participants Who Exhibit a Hematopoietic Response
Description: Hematopoietic response was defined as Hemoglobin (Hb) increment of 2.0 g/dL from baseline or achievement of Hb >= 11 g/dL (whichever occurs first) in the absence of red blood cell transfusions during the preceding 28 days during the treatment period.
Time Frame: 16 Weeks
Measure: Number; unit: Participants
Arm/Group | DA + IV Iron | DA + Oral Iron | DA + Placebo
Number analyzed (Participants) | 164 | 163 | 163
Participants
  Yes | 114 | 109 | 106
  No | 50 | 54 | 57
Statistical Analysis 1: Comparison: DA + IV Iron vs DA + Placebo; With 176 evaluable participants per treatment arm, there would have been >=80% power to detect a difference across two treatment arms of 15% in the primary hematopoietic response endpoint through Fisher's exact test, if the true percentage of patients that experience a hematopoietic response was at least 30% in the superior group, with a 2.5% type I error rate; Test type: Superiority or Other; p = 0.39, Fisher Exact
Statistical Analysis 2: Comparison: DA + Oral Iron vs DA + Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.73, Fisher Exact

2. Secondary Outcome: Percentage of Patients Maintaining an Average Hemoglobin Level Within the National Comprehensive Cancer Network (NCCN) Range (11-13 g/dL) Through Week 16, Once Achieving a Hemoglobin of ≥ 11 g/dL
Time Frame: 16 Weeks
Measure: Number; unit: Percentage of Participants
Arm/Group | DA + IV Iron | DA + Oral Iron | DA + Placebo
Number analyzed (Participants) | 164 | 163 | 163
Percentage of Participants | 10 | 12 | 11

3. Secondary Outcome: Incidence of Patients Receiving at Least One Red Blood Cell (RBC) Transfusions
Time Frame: Week 1 to Week 16
Measure: Number; unit: Participants
Arm/Group | DA + IV Iron | DA + Oral Iron | DA + Placebo
Number analyzed (Participants) | 164 | 163 | 163
Participants
  Yes | 20 | 21 | 22
  No | 144 | 142 | 141
Statistical Analysis 1: Comparison: DA + IV Iron vs DA + Placebo; With 176 evaluable participants per treatment arm, there would have been >=80% power to detect a difference across two treatment arms of 15% in the true percentage of patients that need transfusion was at least 30% in the superior group, with a 2.5% type I error rate; Test type: Superiority or Other; p = 0.7250, Fisher Exact
Statistical Analysis 2: Comparison: DA + Oral Iron vs DA + Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.8700, Fisher Exact

4. Secondary Outcome: Mean Increment in Hemoglobin Level at Week 7
Description: Value at 7 weeks minus value at baseline.
Time Frame: Baseline and 7 weeks
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | DA + IV Iron | DA + Oral Iron | DA + Placebo
Number analyzed (Participants) | 164 | 163 | 163
g/dL | 1.3 (1.35) | 1.1 (1.37) | 1.2 (1.35)
Statistical Analysis 1: Comparison: DA + IV Iron vs DA + Placebo; With 176 evaluable participants per treatment arm, there would have been >=80% power to detect a difference across two treatment arms of 33% of the standard deviation in average hemoglobin levels through two-sided alternative, with a 2.5% type I error rate; Test type: Superiority or Other; p = 0.6639, t-test, 2 sided
Statistical Analysis 2: Comparison: DA + Oral Iron vs DA + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.5660, t-test, 2 sided

5. Secondary Outcome: Mean Increment in Hemoglobin Level at Week 16
Description: Value at 16 weeks minus value at baseline.
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | DA + IV Iron | DA + Oral Iron | DA + Placebo
Number analyzed (Participants) | 164 | 163 | 163
g/dL | 2.1 (1.46) | 2.0 (1.61) | 1.7 (1.64)
Statistical Analysis 1: Comparison: DA + IV Iron vs DA + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.1124, t-test, 2 sided
Statistical Analysis 2: Comparison: DA + Oral Iron vs DA + Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.2051, t-test, 2 sided

6. Secondary Outcome: Time to Hematopoietic Response
Description: Hematopoietic response was defined as Hb increment of 2.0 g/dL from baseline or achievement of Hb >= 11 g/dL (whichever occurs first) in the absence of red blood cell transfusions during the preceding 28 days during the treatment period.
Time Frame: 16 weeks
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | DA + IV Iron | DA + Oral Iron | DA + Placebo
Number analyzed (Participants) | 164 | 163 | 163
Days | 43 [36 to 55] | 61 [55 to 73] | 50 [42 to 64]
Statistical Analysis 1: Comparison: DA + IV Iron vs DA + Oral Iron vs DA + Placebo; Test type: Superiority or Other; p = 0.0648, Log Rank

7. Secondary Outcome: Time to First Red Blood Cell (RBC) Transfusions
Time Frame: 16 weeks
Population: Only 63 participants (20 DA + IV Iron, 21 DA + Oral Iron and 22 DA + Placebo) needed RBC transfusion during 16 weeks of treatment period. Thus, median of time to first RBC transfusion and 95 % confidence interval are not attainable.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | DA + IV Iron | DA + Oral Iron | DA + Placebo
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Change From Baseline in Overall Quality of Life (QOL) Score as Measured by the Linear Analogue Self Assessment (LASA)
Description: Overall QOL item score range: 0 (Worst) to 10 (Best), ordinal. Change: score at 16 weeks minus score at baseline.
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | DA + IV Iron | DA + Oral Iron | DA + Placebo
Number analyzed (Participants) | 164 | 163 | 163
Scores on a scale | 0.4 (2.18) | 0.2 (2.23) | 0.5 (2.28)
Statistical Analysis 1: Comparison: DA + IV Iron vs DA + Placebo; With 176 evaluable participants per treatment arm, there would have been >=80% power to detect a difference across two treatment arms of 33% of the standard deviation in participant QOL through t-test/Wilcoxon test, with a 2.5% type I error rate. A 10 points shift on a 0-100 point scale in QOL measures is generally considered clinically relevant and specifically important in the use of UNISCALE, BFI and FACT-An; Test type: Superiority or Other; p = 0.61, t-test, 2 sided
Statistical Analysis 2: Comparison: DA + Oral Iron vs DA + Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.44, t-test, 2 sided

9. Secondary Outcome: Change From Baseline in Quality of Life (QOL) Score as Measured by Symptom Distress Scale (SDS) at End of Study
Description: SDS Scale range: 0 (Worst), 100 (Best), ordinal. Change: score at 16 weeks minus score at baseline. A clinically significant result will be defined as a shift of 10 points on a 0-100 point transformed scale between the average QOL scores of the 3 variants of iron therapy.
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | DA + IV Iron | DA + Oral Iron | DA + Placebo
Number analyzed (Participants) | 164 | 163 | 163
Scores on a scale | 6.0 (11.73) | 3.5 (11.54) | 5.4 (10.50)
Statistical Analysis 1: Comparison: DA + IV Iron vs DA + Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.62, t-test, 2 sided
Statistical Analysis 2: Comparison: DA + Oral Iron vs DA + Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.30, t-test, 2 sided

10. Secondary Outcome: Change From Baseline in Quality of Life (QOL) Score as Measured by Brief Fatigue Inventory(BFI) Fatigue Now Scale at End of Study
Description: Fatigue Now Scale range: 0 (No Fatigue) to 10 (Worst), ordinal. Change: score at 16 weeks minus score at baseline.
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | DA + IV Iron | DA + Oral Iron | DA + Placebo
Number analyzed (Participants) | 164 | 163 | 163
Scores on a scale | -1.1 (3.08) | -1.1 (2.95) | -1.6 (2.82)
Statistical Analysis 1: Comparison: DA + IV Iron vs DA + Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.19, t-test, 2 sided
Statistical Analysis 2: Comparison: DA + Oral Iron vs DA + Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.17, t-test, 2 sided

11. Secondary Outcome: Change From Baseline in Quality of Life (QOL) Score as Measured by The Functional Assessment of Cancer Therapy-Anemia (FACT-An) at End of Study
Description: FACT-AN Scale range: 0 (Worst) to 100 (Best), ordinal. Change: score at 16 weeks minus score at baseline. A clinically significant result will be defined as a shift of 10 points on a 0-100 point transformed scale between the average QOL scores of the 3 variants of iron therapy.
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | DA + IV Iron | DA + Oral Iron | DA + Placebo
Number analyzed (Participants) | 164 | 163 | 163
Scores on a scale | 8.1 (16.57) | 8.9 (18.97) | 9.5 (18.79)
Statistical Analysis 1: Comparison: DA + IV Iron vs DA + Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.73, t-test, 2 sided
Statistical Analysis 2: Comparison: DA + Oral Iron vs DA + Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.83, t-test, 2 sided

12. Secondary Outcome: C-reactive Protein (CRP) Level at Week 1, Week 7 and Week 16
Time Frame: 1 Week, 7 Weeks and 16 Weeks
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | DA + IV Iron | DA + Oral Iron | DA + Placebo
Number analyzed (Participants) | 164 | 163 | 163
mg/L
  Week 1 | 24.8 (38.12) | 25.4 (36.36) | 31.6 (58.68)
  Week 7 | 28.6 (51.09) | 16.6 (25.25) | 27.0 (49.20)
  Week 16 | 25.6 (46.30) | 16.7 (36.98) | 21.2 (39.07)
Statistical Analysis 1: Comparison: DA + IV Iron vs DA + Oral Iron vs DA + Placebo; Test type: Superiority or Other; p = 0.3852, Kruskal-Wallis — Test Comparison for Week 1 Level
Statistical Analysis 2: Comparison: DA + IV Iron vs DA + Oral Iron vs DA + Placebo; Test type: Superiority or Other; p = 0.0663, Kruskal-Wallis — Test Comparison for Week 7 Level
Statistical Analysis 3: Comparison: DA + IV Iron vs DA + Oral Iron vs DA + Placebo; Test type: Superiority or Other; p = 0.3220, Kruskal-Wallis — Test Comparison for Week 16 Level

13. Secondary Outcome: Soluble Transferrin Receptor (sTfR)Level at Week 1, Week 7 and Week 16
Time Frame: 1 week, 7 weeks and 16 weeks
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | DA + IV Iron | DA + Oral Iron | DA + Placebo
Number analyzed (Participants) | 164 | 163 | 163
mg/L
  Week 1 | 3.9 (2.14) | 4.0 (1.99) | 4.5 (4.52)
  Week 7 | 6.1 (3.04) | 6.2 (2.4) | 7.1 (2.92)
  Week 16 | 5.1 (3.07) | 5.2 (2.19) | 5.6 (2.6)
Statistical Analysis 1: Comparison: DA + IV Iron vs DA + Oral Iron vs DA + Placebo; Test type: Superiority or Other; p = 0.1826, Kruskal-Wallis — Test Comparison for Week 1 Level
Statistical Analysis 2: Comparison: DA + IV Iron vs DA + Oral Iron vs DA + Placebo; Test type: Superiority or Other; p = 0.0113, Kruskal-Wallis — Test comparison for week 7 level
Statistical Analysis 3: Comparison: DA + IV Iron vs DA + Oral Iron vs DA + Placebo; Test type: Superiority or Other; p = 0.3358, Kruskal-Wallis — Test Comparison for week 16 level

14. Secondary Outcome: Ferritin Level at Baseline, Week 7 and Week 16
Time Frame: Baseline, 7 weeks and 16 weeks
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | DA + IV Iron | DA + Oral Iron | DA + Placebo
Number analyzed (Participants) | 164 | 163 | 163
µg/L
  Baseline | 460.5 (526.99) | 479.5 (484.15) | 456.0 (479.27)
  Week 7 | 699.1 (645.31) | 420.6 (498.24) | 478.4 (607.89)
  Week 16 | 726.0 (1037.43) | 425.9 (717.43) | 371.5 (479.87)
Statistical Analysis 1: Comparison: DA + IV Iron vs DA + Oral Iron vs DA + Placebo; Test type: Superiority or Other; p = 0.9022, Kruskal-Wallis — Test comparison for Baseline level
Statistical Analysis 2: Comparison: DA + IV Iron vs DA + Oral Iron vs DA + Placebo; Test type: Superiority or Other; p = 0.0002, Kruskal-Wallis — Test Comparison for Week 7 Level
Statistical Analysis 3: Comparison: DA + IV Iron vs DA + Oral Iron vs DA + Placebo; Test type: Superiority or Other; p = 0.0022, Kruskal-Wallis — Test Comparison for Week 16 Level

15. Secondary Outcome: Mean Corpuscular Volume (MCV) Level at Baseline, Week 7 and Week 16
Description: MCV is a measure of the average red blood cell volume.
Time Frame: Baseline, 7 weeks and 16 weeks
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | DA + IV Iron | DA + Oral Iron | DA + Placebo
Number analyzed (Participants) | 164 | 163 | 163
fL
  Baseline | 90.0 (5.92) | 88.5 (9.05) | 90.1 (8.19)
  Week 7 | 93.0 (9.21) | 92.3 (9.70) | 92.8 (8.56)
  Week 16 | 94.0 (11.37) | 94.4 (7.55) | 92.3 (9.31)
Statistical Analysis 1: Comparison: DA + IV Iron vs DA + Oral Iron vs DA + Placebo; Test type: Superiority or Other; p = 0.1137, Kruskal-Wallis — Test comparison for baseline level
Statistical Analysis 2: Comparison: DA + IV Iron vs DA + Oral Iron vs DA + Placebo; Test type: Superiority or Other; p = 0.8042, Kruskal-Wallis — Test comparison for week 7 level
Statistical Analysis 3: Comparison: DA + IV Iron vs DA + Oral Iron vs DA + Placebo; Test type: Superiority or Other; p = 0.2016, Kruskal-Wallis — Test comparison for week 16 level

16. Secondary Outcome: Transferrin Saturation at Baseline, Week 7 and Week 16
Time Frame: Baseline, 7 weeks and 16 weeks
Measure: Mean (Standard Deviation); unit: Percentage Saturation
Arm/Group | DA + IV Iron | DA + Oral Iron | DA + Placebo
Number analyzed (Participants) | 164 | 163 | 163
Percentage Saturation
  Baseline | 22.5 (12.81) | 19.6 (11.7) | 22.2 (13.36)
  Week 7 | 25.6 (17.48) | 26.4 (23.56) | 21.2 (13.12)
  Week 16 | 26.9 (14.16) | 27.6 (17.81) | 23.9 (15.54)
Statistical Analysis 1: Comparison: DA + IV Iron vs DA + Oral Iron vs DA + Placebo; Test type: Superiority or Other; p = 0.1139, Kruskal-Wallis — Test comparison for baseline level
Statistical Analysis 2: Comparison: DA + IV Iron vs DA + Oral Iron vs DA + Placebo; Test type: Superiority or Other; p = 0.0424, Kruskal-Wallis — Test comparison for week 7 level
Statistical Analysis 3: Comparison: DA + IV Iron vs DA + Oral Iron vs DA + Placebo; Test type: Superiority or Other; p = 0.2025, Kruskal-Wallis — Test comparison for week 16 level

ADVERSE EVENTS:
Arm/Group | DA + IV Iron | DA + Oral Iron | DA + Placebo
Serious Adverse Events (participants affected / at risk) | 5/164 | 3/163 | 2/163
Other Adverse Events (participants affected / at risk) | 150/164 | 147/163 | 141/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DA + IV Iron (N=164) | DA + Oral Iron (N=163) | DA + Placebo (N=163)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Fistula-intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Syndromes (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Investigations) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Investigations) | 2 (2) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DA + IV Iron (N=164) | DA + Oral Iron (N=163) | DA + Placebo (N=163)
Anemia (Blood and lymphatic system disorders) | 6 (9) | 13 (14) | 8 (9)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 2 (4)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Ischemia/Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Restrictive cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Right ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Valvular heart disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Extraocular muscle disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Ocular weakness (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vision-Blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anus Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colonic hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 76 (163) | 72 (166) | 79 (182)
Diarrhea-No Colostom (Gastrointestinal disorders) | 64 (131) | 64 (129) | 68 (131)
Dyspepsia (Gastrointestinal disorders) | 3 (4) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 76 (165) | 83 (164) | 82 (171)
Oral cavity Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2)
Pain-Abdominal (Gastrointestinal disorders) | 3 (3) | 5 (5) | 6 (6)
Pain-Stomach (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Small intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 41 (69) | 37 (70) | 36 (57)
Disease Progression (General disorders) | 5 (5) | 4 (4) | 1 (1)
Edema: Limb (General disorders) | 0 (0) | 1 (2) | 0 (0)
Edema: Viscera (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 20 (32) | 17 (26) | 18 (27)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 3 (3) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Anal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bladder (urinary) infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Bladder infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Blood Infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Bronchus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Colon infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Lung (pneumonia) infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 3 (3) | 3 (3)
Rectum infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Salivary gland infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Skin (cellulites) infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 3 (5) | 1 (1) | 2 (4)
Upper airway infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (2) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (2)
Alkaline phosphatase (Investigations) | 1 (1) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 2 (2)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0) | 3 (3)
CPK (creatine phosphokinase) (Investigations) | 0 (0) | 0 (0) | 1 (1)
Creatinine (Investigations) | 0 (0) | 3 (4) | 2 (2)
Leukopenia (Investigations) | 13 (19) | 17 (25) | 28 (52)
Lymphopenia (Investigations) | 9 (16) | 11 (22) | 10 (22)
Neutropenia (Investigations) | 17 (24) | 17 (21) | 21 (37)
Platelet count decreased (Investigations) | 9 (13) | 15 (23) | 14 (24)
Prothrombin Time (Investigations) | 2 (5) | 0 (0) | 2 (2)
Weight gain (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 5 (6) | 3 (8) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 11 (12) | 8 (9) | 7 (7)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3) | 10 (16) | 6 (7)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 7 (8) | 4 (4) | 5 (7)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 5 (5) | 3 (4) | 4 (6)
Iron increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (4) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (5) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Extremity-lower weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2) | 2 (2)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2)
Trunk weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain-Anal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Ischemia-Cerebral (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Mental status changes (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0)
Neuro (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (8) | 2 (2) | 4 (6)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 4 (4) | 1 (1) | 3 (3)
Syncope Vasovagal (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Glomerular filtration rate (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vaginal fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Adult respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 13 (21) | 8 (9) | 16 (19)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 2 (2) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (4)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 44 (77) | 48 (91) | 46 (77)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 34 (66) | 30 (55) | 33 (58)
Hypertension (Vascular disorders) | 17 (28) | 20 (29) | 14 (16)
Hypotension (Vascular disorders) | 23 (34) | 13 (19) | 24 (31)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 7 (7) | 0 (0) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes